CLINICAL TRIAL: NCT04381338
Title: Pulmonary and Motor Rehabilitation for People With COVID-19 in Intensive Care Units to Reduce Length of Stay in Hospital
Brief Title: Rehabilitation for People With COVID-19 in ICU
Acronym: COVID_REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Prof. S Masiero, University of Padova, Italy (Unknown); Dr. A. Venturin, General Hosipital, Padova, Italy (Unknown); Dr. I. Tiberio, General Hospital, Padova, Italy (Unknown); Dr. D. Zampieri, University of Padova, Italy (Unknown); Dr.ssa M Cattelan, University of Padova, Italy (Unknown); Prof. P. Zanatta, University Hosiptal, Verona, Italy (Unknown); Dr.ssa C. Carollo, General Hospital, Padova, Italy (Unknown); Prof. E. Polati, University Hospital, Verona, Italy (Unknown); Prof. K. Donadello, University Hospital, Verona, Italy (Unknown)
Responsible Party: Principal Investigator, Alessandra Del Felice, MD, PhD, University of Padova
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPadova_1
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Corona Virus Disease 19 (COVID-19); COVID; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Critical Illness
Keywords: Recovery; Outcome; retraining; corona virus disease 19
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Respiratory Distress Syndrome; Critical Illness

STUDY DESIGN:
Intervention Model Description: Clustered, due to catchment area of Hospital with no chance of contamination because of lock down in the area.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation in COVID-19 patients in ICU (Experimental): Every person admitted to ICU for ARDS with a confirmed diagnosis of COVID-19 Motor program
  * Intubated patient GCS >8: passive mobilization; postural positioning GCS< 8: passive and active-assist mobilization; postural positioning
  * Extubated patient
    * If strength < 3 MRC: passive and/or active-assist; functional retraining
    * If strength ≥3 MRC: active-assist and active; strength training; functional retraining Pulmonary Rehabilitation
  * Intubated patient GCS >8: postural positioning GCS< 8: postural positioning, cautious inspiratory muscle training
  * Extubated patient
    * If strength < 3 MRC: postural positioning, positive pressure expiration exercise,inspiratory muscle training
    * If strength ≥3 MRC: postural positioning, positive pressure expiration exercise, inspiratory muscle training The intensity of exercise will prescribed based on the results of the PFIT. and modified Borg Scale.
  Frequency of sessions: 3×15 min/day
  Interventions: Other: Pulmonary and Motor Rehabilitation
- COVID-19 in ICU without Rehabilitation (No Intervention): Standard of care without rehabilitation in ICU

INTERVENTIONS:
Other: Pulmonary and Motor Rehabilitation — Pulmonary and Motor Rehabilitation in ICU
  Arms: Rehabilitation in COVID-19 patients in ICU

SUMMARY:
COVID-19 DISEASE Coronavirus disease 2019 (COVID-19) is a respiratory tract infection caused by a newly emergent coronavirus, severe acute respiratory syndrome from COVID-19, that was first recognized in Wuhan, China, in December 2019. While most people with COVID-19 develop mild or uncomplicated illness, approximately 14% develop severe disease requiring hospitalization and oxygen support and 5% require admission to an intensive care unit. In severe cases, COVID-19 can be complicated by acute respiratory disease syndrome (ARDS) requiring prolonged mechanical ventilation, sepsis and septic shock, multiorgan failure, including acute kidney, liver and cardiac injury.

ARDS REHABILITATION Critically ill people who undergo prolonged mechanical ventilation often develop weakness, with severe symmetrical weakness of and deconditioning of the proximal musculature and of the respiratory muscles (critical illness neuropathy/myopathy).These individuals also develop significant functional impairment and reduced health-related quality of life (HRQL) up to 2 and 5 years after discharge.

ARDS survivors may complain of depression, anxiety, memory disturbances, and difficulty with concentration often unchanged at 2 and 5 years. Less than half of all ARDS survivors return to work within the first year following discharge, two-thirds at two years, and more than 70% at five years.

Early physiotherapy (PT) of people with ARDS has recently been suggested as a complementary therapeutic tool to improve early and late outcomes. The aims of PT programs should be to reduce complications of immobilization and ventilator-dependency, to improve residual function, to prevent new hospitalisations, and to improve health status and HRQL. Physiotherapy in critical patients is claimed also to prevent and contribute to treat respiratory complications such as secretion retention, atelectasis, and pneumonia. Early mobilization and maintenance of muscle strength may reduce the risk of difficult weaning, limited mobility, and ventilator dependency.

Lastly, pulmonary rehabilitation in ICU in mechanically ventilated subjects may reduce length of stay in ICU up to 4.5 day, shorten mechanical ventilation of 2.3 days and weaning by 1.7 days.

The aim of this study is to investigate how early pulmonary and motor rehabilitation impacts on length of hospital admission (ICU and acute ward) and early and late outcomes inpatients that develop ARDS due to COVID-19.

DETAILED DESCRIPTION:
People that develop ARDS due to COVID-19 and requiring admission to ICU (both invasive and non-invasive mechanical ventilation) will be enrolled. Two tertiary referral centers, part of the same region (Veneto) but located in different cities, will recruit participants. ICU standard of care is the same as defined by regional and national guidelines; rehabilitation in ICU COVID-19 subjects is provided only in one center due to local technical and organizational limitations. Non contamination between centers is possible due to restrictions of mobility and strict admission criteria based on catchment area.

Early physiotherapy treatment will start from the day of admission. Baseline measurement of physical function will performed using the Physical Function in ICU Test (PFIT). The PFIT is a submaximal exercise test that was developed for patients in the ICU who may not be able to mobilize away from the bedside.

Participants will start rehabilitation if they will not experiment one of the following conditions or should cease exercise because of the following (see exclusion criteria).

Rehabilitation Intervention

Rehabilitation program will start at admission in ICU. The program is based on the clinical characteristics of the individual to be treated. Participants will commence a hierarchical, standardized protocol that includes functional, respiratory and strength training. If participants will be unable to sit out of bed, assisted active exercises will be performed in bed. Exercise training will be provided for 15 minutes 3 times/day, 6 days per week.

Intensity of strength training: Until fatigue (Borg Scale) Type of strength training: >Grade 3 Medical Research Council (MRC) strength, active to resisted; <Grade 3 MRC strength, active assist to active Repetitions for strength training: Start 5 repetitions each limb, Progress to 3 sets of 10 repetitions as able Functional retraining: Sit-to-stand (using tilt table or standing walker if unable), rolling, supine to sitting, trunk control/balance

Motor program

* Intubated patient Glasgow Coma Scale (GCS) >8: passive mobilisation; postural positioning Glasgow Coma Scale < 8 (weaning): passive and active-assist mobilisation; postural positioning
* Weaned off patient Non-invasively ventilated/O2 high fluxes

  * If strength < 3 MRC: passive and/or active-assist; tentative functional retraining
  * If strength ≥3 MRC: active-assist and active; strength training; functional retraining Pulmonary Rehabilitation
* Intubated patient Glasgow Coma Scale >8: postural positioning Glasgow Coma Scale < 8 (weaning): postural positioning, cautious inspiratory muscle training
* Weaned off patient Non-invasively ventilated/O2 high fluxes

  * If strength < 3 MRC: postural positioning, positive pressure expiration exercise, cautious inspiratory muscle training
  * If strength ≥3 MRC: postural positioning, positive pressure expiration exercise, inspiratory muscle training

The intensity of exercise will prescribed based on the results of the PFIT. Rehabilitation programs will individualized for each patient. Programs will progressed using rates of perceived exertion (RPE) of the modified Borg Scale.

Total session time composition:15 min to complete:

* Whole-body bed exercises + strength + functional retraining
* respiratory rehabilitation Frequency of sessions: 3×15 min/day

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 diagnosis, admitted to ICU with ARDS

Exclusion Criteria:

* Neuromuscular disease, severe heart failure (class IV), persistent severe hypotension (systolic BP < 90mmHg), disorder of consciousness (DoC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Length of ICU stay | up to 60 days
  days of ICU stay

SECONDARY OUTCOMES:
Length of hospital stay | up to 90 days
  days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Del Felice, MD, PhD, Principal Investigator — University of Padova
Locations (2):
- Italy (2):
  - Teaching Hospital, University of Padova, Padua
  - Teaching Hospital, University of Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Bednarik J, Vondracek P, Dusek L, Moravcova E, Cundrle I. Risk factors for critical illness polyneuromyopathy. J Neurol. 2005 Mar;252(3):343-51. doi: 10.1007/s00415-005-0654-x. Epub 2005 Mar 30. PMID 15791390
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Background] Griffiths RD, Hall JB. Intensive care unit-acquired weakness. Crit Care Med. 2010 Mar;38(3):779-87. doi: 10.1097/CCM.0b013e3181cc4b53. PMID 20048676
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Cheung AM, Tansey CM, Tomlinson G, Diaz-Granados N, Matte A, Barr A, Mehta S, Mazer CD, Guest CB, Stewart TE, Al-Saidi F, Cooper AB, Cook D, Slutsky AS, Herridge MS. Two-year outcomes, health care use, and costs of survivors of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):538-44. doi: 10.1164/rccm.200505-693OC. Epub 2006 Jun 8. PMID 16763220
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Adhikari NKJ, Tansey CM, McAndrews MP, Matte A, Pinto R, Cheung AM, Diaz-Granados N, Herridge MS. Self-reported depressive symptoms and memory complaints in survivors five years after ARDS. Chest. 2011 Dec;140(6):1484-1493. doi: 10.1378/chest.11-1667. Epub 2011 Oct 13. PMID 21998261
- [Background] Bienvenu OJ, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Shanholtz C, Husain N, Dennison CR, Herridge MS, Pronovost PJ, Needham DM. Depressive symptoms and impaired physical function after acute lung injury: a 2-year longitudinal study. Am J Respir Crit Care Med. 2012 Mar 1;185(5):517-24. doi: 10.1164/rccm.201103-0503OC. Epub 2011 Dec 8. PMID 22161158
- [Background] Barnato AE, Albert SM, Angus DC, Lave JR, Degenholtz HB. Disability among elderly survivors of mechanical ventilation. Am J Respir Crit Care Med. 2011 Apr 15;183(8):1037-42. doi: 10.1164/rccm.201002-0301OC. Epub 2010 Nov 5. PMID 21057004
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Kress JP, Herridge MS. Medical and economic implications of physical disability of survivorship. Semin Respir Crit Care Med. 2012 Aug;33(4):339-47. doi: 10.1055/s-0032-1321983. Epub 2012 Aug 8. PMID 22875379
- [Background] Ambrosino N, Makhabah DN. Comprehensive physiotherapy management in ARDS. Minerva Anestesiol. 2013 May;79(5):554-63. Epub 2013 Jan 10. PMID 23306398
- [Background] Condessa RL, Brauner JS, Saul AL, Baptista M, Silva AC, Vieira SR. Inspiratory muscle training did not accelerate weaning from mechanical ventilation but did improve tidal volume and maximal respiratory pressures: a randomised trial. J Physiother. 2013 Jun;59(2):101-7. doi: 10.1016/S1836-9553(13)70162-0. PMID 23663795
- [Background] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346
- [Background] Elkins M, Dentice R. Inspiratory muscle training facilitates weaning from mechanical ventilation among patients in the intensive care unit: a systematic review. J Physiother. 2015 Jul;61(3):125-34. doi: 10.1016/j.jphys.2015.05.016. Epub 2015 Jun 16. PMID 26092389
- [Background] Skinner EH, Berney S, Warrillow S, Denehy L. Development of a physical function outcome measure (PFIT) and a pilot exercise training protocol for use in intensive care. Crit Care Resusc. 2009 Jun;11(2):110-5. PMID 19485874
- [Background] Berney S, Haines K, Skinner EH, Denehy L. Safety and feasibility of an exercise prescription approach to rehabilitation across the continuum of care for survivors of critical illness. Phys Ther. 2012 Dec;92(12):1524-35. doi: 10.2522/ptj.20110406. Epub 2012 Aug 9. PMID 22879441
- [Background] Borg G. Ratings of perceived exertion and heart rates during short-term cycle exercise and their use in a new cycling strength test. Int J Sports Med. 1982 Aug;3(3):153-8. doi: 10.1055/s-2008-1026080. PMID 7129724